CLINICAL TRIAL: NCT00051896
Title: Double-Blind, Placebo-Controlled, Dose Escalating, Safety and Pharmacology Study With Three Dosages of GBR 12909 in Cocaine Experienced Volunteers
Brief Title: Assessment of the Potential Interactions Between Cocaine and GBR 12909 - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CPU-0002-1
Record Dates: First submitted 2003-01-17; First posted 2003-01-20 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2005-03

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — vanoxerine

INTERVENTIONS:
Drug: GBR 12909

SUMMARY:
The purpose of this study is to assess the potential interactions between iv cocaine and GBR 12909.

DETAILED DESCRIPTION:
This is a single dose with escalation, double-blind, placebo-controlled inpatient study in which 24 cocaine experienced volunteers that meet protocol eligibility criteria during a 30 day screen period will be randomized into three dose groups.

ELIGIBILITY:
Inclusion Criteria:

* Must understand study procedures and provide written informed consent
* For additional inclusion criteria information, please contact study site for more information.

Exclusion Criteria:

* Please contact study site for more information.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24
Dates: Start 2002-08

PRIMARY OUTCOMES:
Pharmacokinetic parameter comparison

CONTACTS AND LOCATIONS:
Overall Officials: Louis Cantilena, M.D., Principal Investigator — Uniformed Services University of Health Science
Locations (1):
- Uniformed Services University of Health Science, Bethesda, Maryland, United States